CLINICAL TRIAL: NCT03467893
Title: Evaluation of Rebound Effect After Withdrawal of Proton Pump Inhibitor After 8 Weeks of Treatment in Geriatric Population
Brief Title: Evaluation of Rebound Effect After Withdrawal of Proton Pump Inhibitor in Geriatric Population
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EGERIPP
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2018-03

CONDITIONS: Proton Pump Inhibitor
MeSH Terms: interventions — Antacids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antacids — number aof antacids treatment after PPI stop

SUMMARY:
Proton pump inhibitor are frequently used and are short term well tolerated ; but few studies show there are adverse event in long term prescription like fracture or pulmonary infection to Clostridum difficile. The fact is that multi medication in old patient increase the iatrogenic risk and decrease the medication compliance. The Proton pump inhibitor (PPI)are overused in this patient category.Several studies suggest the existence of a rebound effect when people were treated more than 8 weeks ; this effect seems to appear around 14 days after with hyperacidity symptoms.

But there are no studies about old patient. So in this context the aim of the study is to evaluate the prevalence of rebound effect occurence after the end of PPI 8 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in post acute and rehabilitation service
* more than 65 years old
* PPI prescription more than 8 weeks

Exclusion Criteria:

* PPI prescription under 8 weeks
* PPI prescription for digestive haemorragy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient admitted in Leopold Bellan post acute an rehabilitation institution.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Number of antacids used | Day 14 after end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France